CLINICAL TRIAL: NCT05365243
Title: A Pilot Study to Evaluate the Use of the AMMA Portable Scalp Cooling System
Brief Title: A Pilot Study to Evaluate the Use of the AMMA Portable Scalp Cooling System From Cooler Heads
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Single-site study, site was unable to participate
Sponsor: Cooler Heads Care Inc. (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WPH 2201
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Alopecia; Chemotherapy-induced Alopecia; Hair Loss; Breast Cancer; Gynecologic Cancer
MeSH Terms: conditions — Alopecia; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Interventional (Experimental): All patients will use AMMA
  Interventions: Device: AMMA Portalbe Scalp Cooling System

INTERVENTIONS:
Device: AMMA Portalbe Scalp Cooling System — AMMA is indicated for use in chemotherapy infusion centers, during transit from the infusion center and at home and is intended for use by patients who are undergoing chemotherapy treatment and who want to reduce the likelihood of chemotherapy-induced alopecia.

SUMMARY:
Eligible patients will be recruited prior to initiation of chemotherapy for any stage breast or gynecologic cancer. Patients will undergo training in the use of the AMMA Portable Scalp Cooling System and will use the device during each of their chemotherapy treatments. Quality of life and experience of use questionnaires will be completed. Scalp photos and an assessment of hair loss will be preformed at enrollment and at the end of study participation.

DETAILED DESCRIPTION:
AMMA is designed to be used by patients in the chemotherapy infusion center, during transport from the infusion center to home, and after arrival at home. Patients will participate in training in AMMA use and will be asked to bring the device to the chemotherapy infusion center for use during each chemotherapy treatment visit. The device will be used for 30 minutes prior to the start of chemotherapy, during chemotherapy and for 2 hours after chemotherapy. Scalp photos will be obtained at baseline and after the last chemotherapy treatment. Patients will be asked to complete the following questionnaires: training evaluation after training is complete; and symptoms from device use, experience with device use and self-assessment of hair loss after each chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female age 21 years or older at the time of signing informed consent.
* Documented pathologic diagnosis of invasive breast or gynecologic cancer, any stage, requiring treatment with a taxane-containing chemotherapy regimen
* Planned start of treatment with taxane-based chemotherapy in the adjuvant, neoadjuvant or advanced setting
* Plan to complete chemotherapy within 6 months of treatment start
* If received prior chemotherapy causing hair loss, >/= 2 years since last chemotherapy dose and complete recovery of hair
* ECOG performance status 0-1
* Willing and able to sign informed consent for study procedures
* Willing and able to participate in all study procedures

Exclusion Criteria:

* Plan to use chemotherapy regimen other than that listed in inclusion criteria, including any anthracycline-based regimen
* Plan to initiate bone marrow ablation chemotherapy
* History of or plan to initiate whole or partial brain or skull irradiation
* Hormone therapy concurrent with current chemotherapy regimen
* Existing or suspected scalp metastases
* History of concomitant diagnosis of: autoimmune disease affecting hair; cryoglobulinemia; untreated iron deficiency with or without anemia; cold agglutination disease; post-traumatic cold dystrophy; untreated or poorly controlled hyper- or hypothyroidism
* Female pattern baldness
* History of persistent chemotherapy-induced alopecia from prior chemotherapy
* Concomitant exposure to investigational agents, drugs, devices or procedures that cause hair loss
* Concomitant other solid tumor or hematologic malignancy in addition to the current diagnosis

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast and gynecologic cancers
Enrollment: 0 (Actual)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Compliance with AMMA use | 6 months
  Patient-reported questionnaire, including yes/no answers and description of the effectiveness and clarity of the training provided
Experience of AMMA use | 6 months
  Patient-reported questionnaire, including questions on a 1 to 4 scale, where 1 is not at all and 4 is very much, regarding ease of product setup and use in the clinic, during the ride home and at home
Symptoms associated with AMMA use | 6 months
  Patient-reported questionnaire, including questions on a 1 to 4 scale, where 1 is not at all and 4 is very much, regarding amount of hair loss and the impact of any hair loss on daily activities

CONTACTS AND LOCATIONS:
Overall Officials: Kate Dilligan, Study Director — Cooler Heads Care Inc.
Locations (1):
- White Plains Hospital, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No